CLINICAL TRIAL: NCT04907396
Title: International Weight Control Registry
Acronym: IWCR
Status: Recruiting | Type: Observational
Sponsor: Tufts University (Other)
Collaborators: University of Alabama at Birmingham (Other); University of Colorado, Denver (Other); University of Kansas Medical Center (Other); Pennington Biomedical Research Center (Other); University of New Hampshire (Other); United States Military Academy West Point (U.S. Federal Agency)
Responsible Party: Principal Investigator, Susan Roberts, Co-Principal Investigator, Tufts University
Other Study IDs: 13075
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Weight Loss; Overweight; Obesity
Keywords: Weight Loss Maintenance; Obesity Management
MeSH Terms: conditions — Weight Loss; Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The IWCR is a global scientific study aimed at better understanding the opportunities and barriers for reducing the prevalence of obesity by collecting information from people who have experience with weight management in their everyday lives. The investigators seek to gather information on a wide range of weight management experiences, ranging from weight loss and weight loss maintenance to weight gain and inability to lose weight.

ELIGIBILITY:
Inclusion Criteria:

* The IWCR is open to anyone 18 years or older who is considering weight loss, is actively engaged in weight loss, or has previously attempted weight loss (including successful and unsuccessful attempts)

Exclusion Criteria:

1. Minors, below the age of 18
2. Adults who are not able to give informed consent online and complete online surveys

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 100,000 participants who meet eligibility requirements
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2020-12-10 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Percent weight change | 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Susan B Roberts, PhD, Principal Investigator — Tufts University; James O Hill, PhD, Principal Investigator — University of Alabama at Birmingham; Sai K Das, PhD, Study Director — Tufts University; Drew Sayer, PhD, Study Director — University of Alabama at Birmingham
Locations (7):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Colorado, Denver, Denver, Colorado
  - University of Kansas Medical Center, Kansas City, Kansas
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts
  - University of New Hampshire, Durham, New Hampshire
  - United States Military Academy, West Point, West Point, New York

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared. Specific to be determined

REFERENCES:
- [Derived] Chui TK, Cedillo YE, El Zein A, Pavela G, Caldwell AE, Peters JC, Friedman JE, DebRoy S, Oslund JL, Das SK, Roberts SB, Hill JO, Sayer RD. Evaluation of socioecological factors on health behaviors and weight change during major life event: A cross-sectional study using data collected during the COVID-19 pandemic. Obes Sci Pract. 2024 Aug 10;10(4):e785. doi: 10.1002/osp4.785. eCollection 2024 Aug. PMID 39130192
- [Derived] Caldwell AE, More KR, Chui TK, Sayer RD. Psychometric validation of four-item exercise identity and healthy-eater identity scales and applications in weight loss maintenance. Int J Behav Nutr Phys Act. 2024 Feb 23;21(1):21. doi: 10.1186/s12966-024-01573-y. PMID 38395833
- [Derived] Roberts SB, Das SK, Sayer RD, Caldwell AE, Wyatt HR, Mehta TS, Gorczyca AM, Oslund JL, Peters JC, Friedman JE, Chiu CY, Greenway FL, Donnelly JE, Dao MC, Cuevas AG, Affuso O, Wilkinson LL, Thomas D, Al-Ozairi E, Yannakoulia M, Khazrai YM, Manalac RJ, Bachiashvili V, Hill JO. Technical report: an online international weight control registry to inform precision approaches to healthy weight management. Int J Obes (Lond). 2022 Sep;46(9):1728-1733. doi: 10.1038/s41366-022-01158-4. Epub 2022 Jun 16. PMID 35710944
- See also: International Weight Control Registry Website — http://internationalweightcontrolregistry.org